CLINICAL TRIAL: NCT06163001
Title: Effects of Supervised Aerobic and Resistance Exercises on Measures of Frailty in Chronic Liver Disease Patients Undergoing Living Donor Liver Transplantation- an Open Label Randomised Controlled Trial
Brief Title: Role of Exercise in Chronic Liver Disease Patients Undergoing Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ILBS-LDLT-02
Record Dates: First submitted 2023-08-28; First posted 2023-12-08 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Chronic Liver Disease and Cirrhosis; Frailty
Keywords: exercise
MeSH Terms: conditions — Fibrosis; Frailty; Motor Activity | interventions — Physical Therapy Modalities; Exercise Therapy; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental)
  Interventions: Behavioral: Supervised aerobic and resistance exercises; Dietary Supplement: Dietary supplementation
- Dietary supplementation (Active Comparator)
  Interventions: Dietary Supplement: Dietary supplementation

INTERVENTIONS:
Behavioral: Supervised aerobic and resistance exercises — 4 weeks of preoperative supervised aerobic and resistance exercises
  Other Names: physiotherapy; exercise therapy
  Arms: Exercise Group
Dietary Supplement: Dietary supplementation — 4 weeks of preoperative Standard medical therapy which will consist of dietary advice and supplementation

SUMMARY:
The goal of this randomised clinical trial (open label) is to test the effect of supervised aerobic and resistance exercises in chronic liver disease patients being planned for living donor liver transplantation (LDLT). The main question it aims to answer are:

* If pre-operative supervised aerobic and resistance exercise for 4 weeks can improve the measures of frailty (Liver frailty index, Short physical performance battery, pulmonary function tests) in chronic liver disease patients being planned for LDLT.
* Can this approach also translate into clinically significant benefits in the postoperative outcomes of LDLT.

Participants will be randomised into two groups receiving either

1. Standard medical therapy along with supervised aerobic and resistance exercises for 4 weeks.
2. Standard medical therapy. The two groups will be compared for progression of the measures of frailty ver the course of their participation as well as their post LDLT outcomes.

DETAILED DESCRIPTION:
1. Aim and Objective - Primary objective: To assess effects of pre-operative aerobic and resistance exercises in decompensated CLD patients planned for LDLT on the measures of frailty after 1 month of supervised exercise.

   Secondary objectives: To assess effects of pre-operative aerobic and resistance exercises in decompensated CLD patients planned for LDLT on the post LDLT outcomes, myostatin levels (on POD 14) and skeletal muscle mass (on POD14).
2. Methodology:

   * Study population - Consecutive voluntary adults (>18 years) with chronic liver disease, planned for living donor liver transplantation fulfilling the conditions as per inclusion and exclusion criteria.
   * Study design - Interventional study- Open label randomised controlled trial
   * Study period - From time of ethical clearance till 31st December 2024
   * Sample size - Assuming median LFI for CLD patients as 3.9 ± 0.3*, and assuming an improvement of 5% with introduction of exercise along with SMT after 1 follow up, and keeping alpha of 5%, and power of study as 90%, with 1:1 ratio of cases and controls, then by method of change we need to enroll a total of 54 patients with 27 in each arm. Assuming 10% non compliance, a total of 60 cases will be enrolled, with 30 cases in each arm.
   * Intervention - Pre-operative supervised exercise-based regimen versus standard medical therapy alone for a minimum duration of 4 weeks.
   * Monitoring and assessment - Clinical profile of the patient and symptoms will be serially followed during the patients OPD visits.
   * Adverse effects - Exercise may aggravate encephalopathy, metabolic disorders, AKI/HRS. It may also lead to falls due to cardio-pulmonary intolerance or hepatic encephalopathy.
   * Stopping rule - Inability to follow the exercise schedule, or development of any of the adverse effects due to exercise as mentioned above.
3. Expected outcome of the project: Better values of measures of frailty and post LDLT outcomes in patients receiving pre-operative concurrent exerises as an intervention.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary adult patient (>18 years), decompensated chronic liver disease patients planned for LDLT, and Who pass the screening tests done in the OPD

  1. Able to follow the introductory level exercises as per the protocol in the OPD without any adverse event.
  2. No drop in the spO2 less than 93% on a 6 minute walk test.

Exclusion Criteria:

1. Patients with a physical disability (upper or lower limb deformity/abnormality)
2. Exercise intolerance or inability to follow exercise regime.
3. Patients who fail the screening tests.
4. Patients on the following drugs-

   * Higher corticosteroid dose (>0.1mg/kg/day),
   * BCAA (Branched chain amino acids)
   * Growth hormone, testosterone, SARMs,
   * Ghrelin agonists, myostatin antibodies,
   * Activin IIR antagonists, angiotensin converting enzyme inhibitors,
   * Espindolol (mixed beta agonist and antagonists), and
   * Fast skeletal muscle troponin activators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Liver frailty index | 4 weeks post intervention, Post op day 14, Post op day 30
  Robust defined as LFI <3.2, prefrail defined as LFI between 3.2 and 4.4, and frail defined as LFI ≥4.5
short physical performance battery | 4 weeks post intervention, Post op day 14, Post op day 30
  SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness
pulmonary function test | 4 weeks post intervention, Post op day 14, Post op day 30
  PEF would be tested
pulmonary function test | 4 weeks post intervention, Post op day 14, Post op day 30
  FEV1 would be tested

SECONDARY OUTCOMES:
Time to extubation | Till Post op day 90
Need for re-intubation | Till Post op day 90
Duration of NIV support | Till Post op day 90
Mortality | 90 days
Myostatin levels in blood | Post intervention at 4 weeks & on Post op day 14
Skeletal muscle mass- L3 Skeletal Muscle Index | Post intervention at 4 weeks & on Post op day 14
Time to mobilization out of bed | Till Post op day 90
Length (Days) of ICU stay | Till Post op day 90
Number of days of hospital stay | Till Post op day 90
Incidence of all septic complications | Till Post op day 90
Major surgical complications (CDC > grade 3) | Till Post op day 90
Pulmonary complications- Clinical evaluation | Till Post op day 90

CONTACTS AND LOCATIONS:
Overall Officials: Viniyendra Pamecha, MS FEBS FRCS(UK), Study Chair — Professor and HOD HPB Surgery and Liver Transplantation
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No